CLINICAL TRIAL: NCT01966653
Title: Randomised Clinical Trial Comparing Fosfomycin vs. Nitrofurantoin for Treatment of Uncomplicated Lower Urinary Tract Infection in Female Adults at Increased Risk of Antibiotic-resistant Bacterial Infection
Brief Title: Study Comparing Nitrofurantoin to Fosfomycin for Acute Urinary Tract Infection in Women
Acronym: AIDA-WP2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Stephen Harbarth, Professor Stephan Harbarth, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-014
Record Dates: First submitted 2013-10-10; First posted 2013-10-21 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Urinary Tract Infections; Cystitis
Keywords: nitrofurantoin; fosfomycin; urinary tract infection; clinical efficacy; bacteriologic response
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — Nitrofurantoin; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitrofurantoin (Active Comparator): Nitrofurantoin will be given orally at a dose of 100 mg three times daily for 5 days.
  Interventions: Drug: nitrofurantoin
- fosfomycin (Active Comparator): A single 3g dose of oral fosfomycin will be given.
  Interventions: Drug: fosfomycin

INTERVENTIONS:
Drug: nitrofurantoin — nitrofurantoin 100 mg po tid for 5 days
  Other Names: Macrodantin; Furadantine
  Arms: nitrofurantoin
Drug: fosfomycin — fosfomycin 3g po single dose
  Other Names: Monuril
  Arms: fosfomycin

SUMMARY:
Developed before the establishment of a structured process for drug assessment, nitrofurantoin is now being prescribed frequently given the rise in multi-resistant gram-negative pathogens. Doubts remain regarding fosfomycin's long-term clinical effectiveness. A randomized, controlled trial is needed to explore the clinical effectiveness and better define the side effect profiles of both nitrofurantoin and fosfomycin. This multi-center open trial will randomize 600 non-pregnant women at three international sites (200 each in Poland, Switzerland, and Israel) at increased risk for carriage of resistant uropathogens and with suspicion of uncomplicated lower urinary tract infection to receive either oral nitrofurantoin 100 mg three times daily for 5 days or a single 3g dose of oral fosfomycin. Patients will be followed for clinical and bacteriologic response at days 14 and 28 post therapy completion. The study hypothesis holds that nitrofurantoin will be superior to fosfomycin in clinical efficacy at final follow-up.

DETAILED DESCRIPTION:
Developed before the establishment of a structured process for drug assessment, nitrofurantoin is now being prescribed frequently given the rise in multi-resistant gram-negative pathogens. Doubts remain regarding fosfomycin's long-term clinical effectiveness. A randomized, controlled trial is needed to explore the clinical effectiveness and better define the side effect profiles of both nitrofurantoin and fosfomycin. From autumn 2013 through summer 2016, this multi-center open trial will randomize 600 non-pregnant women at three international sites (200 each in Poland, Switzerland, and Israel) at increased risk for carriage of resistant uropathogens and with suspicion of uncomplicated lower urinary tract infection to receive either oral nitrofurantoin 100 mg three times daily for 5 days or a single 3g dose of oral fosfomycin. Patients will be followed for clinical and bacteriologic response at days 14 and 28 post therapy completion. The study hypothesis holds that nitrofurantoin will be superior to fosfomycin in clinical efficacy at final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥ 18 years
* Written informed consent
* At least one of four key UTI symptoms that could be attributed to an uncomplicated UTI, and no alternative explanation (i.e. symptoms suggestive of STI or vulvo-vaginitis):
* Dysuria
* Urgency (including nocturia)
* Frequency
* Suprapubic tenderness
* Urine dipstick test positive for either nitrites or leukocyte esterase
* Patient is at increased risk for resistant pathogens, e.g., FQ-resistant or ESBL-producing Enterobacteriacae

Exclusion Criteria:

* Male sex
* Pregnancy or planned pregnancy
* Known carriage of nitrofurantoin- or fosfomycin-resistant uropathogens(s)
* Concomitant antimicrobial therapy
* Use of any antibiotics in the past 7 days
* Known or suspected hypersensitivity or allergy to fosfomycin or nitrofurantoin
* History of lung or liver reaction or peripheral neuropathy after use of nitrofurantoin or other nitrofurans in the past
* Pre-existing polyneuropathy
* G6PD deficiency
* Symptoms consistent with UTI in the preceding 4 weeks
* Active upper UTI (e.g. pyelonephritis, urosepsis: fever > 38.0, flank pain, chills)
* Symptoms/signs suggestive of vaginitis or sexually transmitted infection
* Indwelling catheter, nephrostomy, ureter stent or other foreign material
* Otherwise complicated UTI:
* A history of anatomical or functional abnormalities of the urogenital tract:
* Congenital abnormalities
* Polycystic kidney disease
* Obstruction or stricture of renal pelvis, ureter or urethra
* Kidney stones
* Cystocele
* Cystic diverticulae
* Change of anatomical proportions (e.g. after ureter implantation)
* Chronic vesico-urethral reflux
* Neurogenic bladder
* Severe chronic renal (creatinine clearance < 30 ml/min) or hepatic dysfunction
* Porphyria
* Immunosuppression:
* Untreated infection with the human immunodeficiency virus (HIV)
* Use of high-dose systemic corticosteroids or other immunosuppressive medication
* Chemotherapy
* Treatment with radiation
* Critical illness requiring intensive care
* Planned surgery within the next 6 weeks
* Inability to take oral drugs
* Participation in another prospective clinical trial
* Previous enrolment in the proposed study
* Inability to understand or to follow the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical cure, clinical failure, or indeterminate clinical response (see description below) | at 28 days post therapy completion
  Clinical response is defined as either (1) clinical cure, which in turn is defined as complete resolution of symptoms with no recurrence of symptoms or signs of urinary tract infection; (2) clinical failure, defined as the need for additional, or change in, antibiotic treatment due to a urinary tract infection, OR discontinuation due to lack of efficacy; or (3) indeterminate response, defined as either persistence of symptoms without objective evidence of infection (absence of bacteriuria or pyuria) OR any extenuating circumstances precluding a classification or clinical cure/failure.

SECONDARY OUTCOMES:
Number of participants with bacteriologic cure and with bacteriologic recurrence | at 28 days post therapy completion
  Bacteriologic response is defined as either (1) bacteriologic cure, that is, eradication of the infecting strain with no recurrence of bacteriuria (<10x3 cfu/mL) during follow-up; or (2) bacteriologic recurrence, defined as bacteriuria >10x3 cfu/mL. However, bacteriologic recurrence without urinary tract symptoms will be designated asymptomatic bacteriuria and left untreated.

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | within 28 days post therapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Harbarth, MD, MS, Principal Investigator — University of Geneva
Locations (3):
- Tel Aviv University, Tel Aviv, Israel
- Lodz University Hospital, Lodz, Poland
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Huttner A, Kowalczyk A, Turjeman A, Babich T, Brossier C, Eliakim-Raz N, Kosiek K, Martinez de Tejada B, Roux X, Shiber S, Theuretzbacher U, von Dach E, Yahav D, Leibovici L, Godycki-Cwirko M, Mouton JW, Harbarth S. Effect of 5-Day Nitrofurantoin vs Single-Dose Fosfomycin on Clinical Resolution of Uncomplicated Lower Urinary Tract Infection in Women: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1781-1789. doi: 10.1001/jama.2018.3627. PMID 29710295
- See also: Related info. — http://www.aida-project.eu/